CLINICAL TRIAL: NCT03237156
Title: A Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose, Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of TAK-906 in Japanese Healthy Male Subjects
Brief Title: Phase 1 TAK-906 Single and Multiple Ascending Dose Study in Japanese Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: TAK-906-1004; U1111-1197-9663 (Registry Identifier: WHO); JapicCTI-173661 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2017-07-31; First posted 2017-08-02 (Actual); Results first posted 2019-02-18 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2020-12

CONDITIONS: Japanese Healthy Adult Male Participants
Keywords: Drug therapy
MeSH Terms: interventions — trazpiroben

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- TAK-906 50 mg; Cohort 1 (Experimental): TAK-906 50 milligram (mg) capsules, orally, once daily on Day 1 as Single Dose Period followed by TAK-906 50 mg capsules, orally, twice daily from Day 3 to 7 as Multiple Dose Period.
  Interventions: Drug: TAK-906
- TAK-906 Placebo; Cohort 1 (Placebo Comparator): TAK-906 Placebo capsules, orally, once daily on Day 1 as Single Dose Period followed by TAK-906 Placebo capsules, orally, twice daily from Day 3 to 7 as Multiple Dose Period.
  Interventions: Drug: TAK-906 Placebo
- TAK-906 100 mg; Cohort 2 (Experimental): TAK-906 100 mg capsules, orally, once daily on Day 1 as Single Dose Period followed by TAK-906 100 mg capsules, orally, twice daily from Day 3 to 7 as Multiple Dose Period. Cohort 2 will be conducted after Cohort 1.
  Interventions: Drug: TAK-906
- TAK-906 Placebo; Cohort 2 (Placebo Comparator): TAK-906 Placebo capsules, orally, once daily on Day 1 as Single Dose Period followed by TAK-906 Placebo capsules, orally, twice daily from Day 3 to 7 as Multiple Dose Period. Cohort 2 will be conducted after Cohort 1.
  Interventions: Drug: TAK-906 Placebo
- TAK-906 10 mg; Cohort 3 (Experimental): TAK-906 10 mg capsules, orally, once daily on Day 1 as Single Dose Period followed by TAK-906 10 mg capsules, orally, twice daily from Day 3 to 7 as Multiple Dose Period.
  Interventions: Drug: TAK-906
- TAK-906 Placebo; Cohort 3 (Placebo Comparator): TAK-906 Placebo capsules, orally, once daily on Day 1 as Single Dose Period followed by TAK-906 Placebo capsules, orally, twice daily from Day 3 to 7 as Multiple Dose Period.
  Interventions: Drug: TAK-906 Placebo

INTERVENTIONS:
Drug: TAK-906 — TAK-906 capsules.
  Arms: TAK-906 10 mg; Cohort 3; TAK-906 100 mg; Cohort 2; TAK-906 50 mg; Cohort 1
Drug: TAK-906 Placebo — Placebo capsules.
  Arms: TAK-906 Placebo; Cohort 1; TAK-906 Placebo; Cohort 2; TAK-906 Placebo; Cohort 3

SUMMARY:
The purpose of this study is to evaluate safety, tolerability, pharmacokinetics, and pharmacodynamics of single and multiple oral doses of TAK-906 in Japanese healthy male participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-906. TAK-906 is being tested in healthy participants in order to evaluate safety and tolerability of single and multiple oral doses of TAK-906 in Japanese healthy male participants.

The study will enroll approximately 24 participants. Participants will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups in Cohort 1 or Cohort 3. Study drug will be administered in a double-blind manner which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need), orally, once daily on Day 1 as Single Dose Period and twice daily from Day 3 to 7 as Multiple Dose Period:

* TAK-906 50 mg (Cohort 1)
* TAK-906 100 mg (Cohort 2)
* TAK-906 10 mg (Cohort 3)
* Placebo (dummy inactive pill) - this is a tablet that looks like the study drug but has no active ingredient

Cohort 2 will be conducted after the completion of Cohort 1. This will be conducted in Japan.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator or sub-investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant signs and dates a written, informed consent form prior to the initiation of any study procedures.
3. The participant is a Japanese healthy adult male, aged 20 to 60 years, inclusive, at the time of informed consent.
4. The participant weighs at least 50 kilogram (kg) and has a body mass index (BMI) from 18.5 to 25 kilogram per square meter (kg/m^2), inclusive at Screening.
5. A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from the signing of informed consent to 12 weeks (84 days) after the last dose of study drug. The female partner of a male participant should also be advised to use adequate contraception.

Exclusion Criteria:

1. The participant has received any investigational compound within 16 weeks (112 days) prior to the first dose of study drug.
2. The participant has received TAK-906 in a previous clinical study or as a therapeutic agent.
3. The participant is an immediate family member of or an investigational site employee, or is in a dependent relationship with an investigational site employee who is involved in the conduct of this study (example, spouse, parent, child, sibling) or may consent under duress.
4. The participant has uncontrolled, clinically significant neurologic, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, or endocrine disease or other abnormality, which may impact the ability of the participant to participate in the study or potentially confound its results.
5. The participant has a history of any psychiatric disease that would interfere with the evaluation of study drug activity (prolactin concentration) or safety.
6. The participant has a history of seizure or tardive dyskinesia.
7. The participant has a history of hyperprolactinemia, pituitary adenoma, and/or hypothyroidism.
8. The participant has a family history of prolonged QT.
9. The participant has undergone previous gastric bypass surgery or currently had a gastric band fitted.
10. The participant has dysphagia and/or inability to swallow study medication whole.
11. The participant has a known hypersensitivity to any component of the TAK-906 formulation or related compounds.
12. The participant has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 2 years prior to the Screening visit, or is unwilling to agree to abstain from alcohol and drugs throughout the study, or has a positive urine test result for drugs of abuse or a positive alcohol screen (urine alcohol test/breath test) result for alcohol at Screening.
13. The participant has taken any excluded medication, supplements, or dietary products during the time periods listed in the Excluded Medications, Supplements, and Dietary Products table.
14. If male, the participant intends to donate sperm during the course of this study or for at least 12 weeks (84 days) after the last dose of study drug.
15. The participant has current or recent (within 24 weeks [168 days]) gastrointestinal disease that would be expected to influence the absorption of drugs (that is, a history of malabsorption, esophageal reflux, peptic ulcer disease, erosive esophagitis, frequent [more than once per week] occurrence of heartburn, or any surgical intervention).
16. The participant has a history of cancer, except basal cell carcinoma which has been in remission for at least 5 years prior to Day 1.
17. The participant has a positive test result for hepatitis B virus surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody/antigen, or serological reactions for syphilis at Screening.
18. The participant has used nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patch or nicotine gum) within 4 weeks (28 days) prior to the first dose of study drug. Cotinine test is positive at Screening.
19. The participant has poor peripheral venous access.
20. The participant has undergone whole blood collection of at least 200 mL within 4 weeks (28 days) or at least 400 mL within 12 weeks (84 days) prior to the start of study drug administration.
21. The participant has undergone whole blood collection of at least 800 mL in total within 52 weeks (364 days) prior to the start of study drug administration.
22. The participant has undergone blood component collection within 2 weeks (14 days) prior to the start of study drug administration.
23. The participant has a Screening or Check-in (Day -1) electrocardiogram (ECG) that was abnormal (clinically significant).
24. The participant has a QTcF of greater than (>) 450 millisecond (msec) on the ECG at Screening, at Check-in (Day -1), or prior to the first dose of study drug (Day 1 predose).
25. The participant has abnormal Screening or Day -1 laboratory values that suggest a clinically significant underlying disease or any participant with the following lab abnormalities:

    * Transaminase (alanine aminotransferase [ALT] and/or aspartate aminotransferase [AST]) and/or total bilirubin >1.5 × upper limit of normal (ULN).
    * Creatinine >1.2 milligram per deciliter (mg/dL).
26. The participant who, in the opinion of the investigator or sub-investigator, is unlikely to comply with the protocol or is unsuitable for any other reason.

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2017-10-07 (Actual); Study Completion 2017-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Sekino Clinical Pharmacology Clinic, Toshima City, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in Japan from 07 August 2017 to 07 October 2017.
Pre-assignment Details: Healthy male participants were enrolled in this study to receive TAK-906 as: single ascending dose and multiple ascending dose of 50 milligram (mg) in Cohort 1, 100 mg in Cohort 2, and 10 mg in Cohort 3.
Groups:
- Cohorts 1-3: Placebo: TAK-906 placebo-matching capsule, orally, once on Day 1 in Single Dose Period, followed by TAK-906 placebo-matching capsules, orally twice daily from Day 3 to Day 7 in Multiple Dose Period.
- Cohort 1: TAK-906 50 mg: TAK-906 50 mg, capsule, orally, once on Day 1 in Single Dose Period, followed by TAK-906 50 mg, capsules, orally, twice daily from Day 3 to Day 7 in Multiple Dose Period.
- Cohort 2: TAK-906 100 mg: TAK-906 100 mg, capsule, orally, once on Day 1 in Single Dose Period, followed by TAK-906 100 mg, capsules, orally, twice daily from Day 3 to Day 7 in Multiple Dose Period.
- Cohort 3: TAK-906 10 mg: TAK-906 10 mg, capsule, orally, once on Day 1 in Single Dose Period, followed by TAK-906 10 mg, capsules, orally, twice daily from Day 3 to Day 7 in Multiple Dose Period.
Period: Overall Study
Arm/Group | Cohorts 1-3: Placebo | Cohort 1: TAK-906 50 mg | Cohort 2: TAK-906 100 mg | Cohort 3: TAK-906 10 mg
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The pharmacokinetic (PK) analysis set consisted of participants who received at least 1 dose of the study drug, completed the minimum protocol-specified procedures with no significant protocol deviations, and who were evaluable for the PK.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohorts 1-3: Placebo | Cohort 1: TAK-906 50 mg | Cohort 2: TAK-906 100 mg | Cohort 3: TAK-906 10 mg | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.5 (6.80) | 27.7 (4.68) | 27.8 (8.04) | 29.0 (4.52) | 28.5 (5.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Japan | 6 | 6 | 6 | 6 | 24
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 170.2 (6.11) | 172.0 (2.53) | 172.3 (5.32) | 171.5 (3.89) | 171.5 (4.43)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 63.20 (7.685) | 63.12 (5.221) | 63.17 (6.914) | 66.55 (5.375) | 64.01 (6.139)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 21.80 (2.107) | 21.35 (1.871) | 21.25 (1.819) | 22.63 (1.725) | 21.76 (1.845)
Smoking Classification: Never Smoked [Count of Participants; unit: Participants] | 6 | 6 | 6 | 6 | 24
Consumption of Alcohol [Count of Participants; unit: Participants]
  Had a few times per month | 0 | 2 | 2 | 0 | 4
  Had no alcohol consumption | 6 | 4 | 4 | 6 | 20
Consumption of Caffeine [Count of Participants; unit: Participants]
  Had caffeine consumption | 2 | 4 | 2 | 2 | 10
  Had no caffeine consumption | 4 | 2 | 4 | 4 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experience at Least One Treatment-Emergent Adverse Event (TEAE)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical investigation participant who has signed informed consent to participate in a study; it does not necessarily have to have a causal relationship with the treatment or study participation. A treatment-emergent adverse events (TEAE) is defined as an AE whose date of onset occurs on or after the start of study drug.
Time Frame: Baseline up to Day 14
Population: The safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1-3: Placebo | Cohort 1: TAK-906 50 mg | Cohort 2: TAK-906 100 mg | Cohort 3: TAK-906 10 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 1 | 0 | 2 | 1

2. Primary Outcome: Number of Participants With Markedly Abnormal Values of Vital Signs
Description: Reported data were numbers of participants who met markedly abnormal criteria of vital signs. Vital signs included body temperature, respiratory rate, blood pressure, and pulse. Vital signs collected were classified as markedly abnormal values if they met the following criteria: systolic blood pressure less than (<) 85 millimeter of mercury (mmHg) or greater than (>) 180 mmHg, diastolic blood pressure <50 mmHg or >110 mmHg, pulse <50 beats per minute (bpm) or >120 bpm, body temperature <35.6 °C or >37.7 °C.
Time Frame: Baseline up to Day 14
Population: The safety analysis set included all participants who received at least 1 dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1-3: Placebo | Cohort 1: TAK-906 50 mg | Cohort 2: TAK-906 100 mg | Cohort 3: TAK-906 10 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Diastolic blood pressure <50 mmHg | 2 | 1 | 2 | 1
  Pulse < 50 bpm | 3 | 2 | 2 | 2

3. Primary Outcome: Number of Participants With Markedly Abnormal Values of Clinical Laboratory Test Results
Description: Reported data were numbers of participants who met markedly abnormal criteria of clinical laboratory test results. Clinical laboratory test results collected were classified as markedly abnormal values if they met the following criteria: red blood cells <0.8×lower limit of normal (LLN) or >1.2×upper limit of normal (ULN), platelets <75×10^3/μL or >600×10^3/μL, white blood cells <0.5×LLN or >1.5×ULN, protein (total) <0.8×LLN or >1.2×ULN, albumin <2.5 g/dL, blood urea nitrogen >30 mg/dL, uric acid >13.0 mg/dL, creatinine >2.0 mg/dL, total cholesterol >300 mg/dL, triglycerides >2.5×ULN, bilirubin (total) >2.0 mg/dL, Sodium <130 mEq/L or >150 mEq/L, Potassium <3.0 mEq/L or >6.0 mEq/L, Chloride <75 mEq/L or >126 mEq/L, Calcium <7.0 mg/dL or >11.5 mg/dL, Phosphorus <1.6 mg/dL or >6.2 mg/dL, alkaline phosphatase >3×ULN, aspartate aminotransferase >3×ULN, alanine aminotransferase >3×ULN, gamma-glutamyl transferase >3×ULN, glucose <50 mg/dL or >350 mg/dL, Magnesium <1.2 mg/dL or >3.0 mg/dL.
Time Frame: Baseline up to Day 14
Population: The safety analysis set included all participants who received at least 1 dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1-3: Placebo | Cohort 1: TAK-906 50 mg | Cohort 2: TAK-906 100 mg | Cohort 3: TAK-906 10 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Markedly Abnormal Values of 12-lead Electrocardiogram (ECG)
Description: Reported data were numbers of participants who met markedly abnormal criteria of 12-lead ECG. A standard 12-lead ECG was performed. The data collected was classified as markedly abnormal values if it met the following criteria: heart rate <50 bpm or >120 bpm, QT interval less than or equal to (<=) 50 msec or greater than or equal to (>=) 460 msec, QTcF interval <=50 msec or either of the following conditions was met: observed value >=500 msec, change from Day 1 Predose >= 30 msec and observed value >=450 msec.
Time Frame: Baseline up to Day 8
Population: The safety analysis set included all participants who received at least 1 dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1-3: Placebo | Cohort 1: TAK-906 50 mg | Cohort 2: TAK-906 100 mg | Cohort 3: TAK-906 10 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Heart Rate <50 bpm | 3 | 1 | 3 | 2
  QT Interval >= 460 msec | 1 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With TEAEs Related to Physical Examinations
Description: as for outcome 1
Time Frame: Baseline up to Day 14
Population: The safety analysis set included all participants who received at least 1 dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1-3: Placebo | Cohort 1: TAK-906 50 mg | Cohort 2: TAK-906 100 mg | Cohort 3: TAK-906 10 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0

6. Secondary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-906 and Its Metabolite M23 on Day 1 of Single Dose Period
Description: AUC∞ is a measure of total plasma exposure to TAK-906 and its Metabolite M23 from Time 0 extrapolated to infinity, calculated using the observed value of the last quantifiable concentration.
Time Frame: Day 1 pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours post-dose
Population: The PK analysis set consisted of participants who received at least 1 dose of the study drug, completed the minimum protocol-specified procedures with no significant protocol deviations, and who were evaluable for the PK.
Measure: Geometric Mean (Standard Deviation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Cohort 1: TAK-906 50 mg | Cohort 2: TAK-906 100 mg | Cohort 3: TAK-906 10 mg
Number analyzed (Participants) | 6 | 6 | 6
hour*nanogram per milliliter (h*ng/mL)
  TAK-906 | 72.58 (17.329) | 156.9 (38.048) | 13.71 (2.1631)
  Metabolite M23 | 7.869 (2.1260) | 16.05 (7.5395) | 1.602 (0.46441)

7. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-906 and Its Metabolite M23 on Day 1 of Single Dose Period
Description: Cmax is the peak plasma concentration of TAK-906 and its metabolite M23.
Time Frame: Day 1 pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours post-dose
Population: as for outcome 6
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Cohort 1: TAK-906 50 mg | Cohort 2: TAK-906 100 mg | Cohort 3: TAK-906 10 mg
Number analyzed (Participants) | 6 | 6 | 6
nanogram per milliliter (ng/mL)
  TAK-906 | 35.31 (12.255) | 58.21 (28.491) | 6.951 (2.0380)
  Metabolite M23 | 3.082 (0.63298) | 4.412 (3.0329) | 0.5088 (0.28496)

8. Secondary Outcome: AUCtau: Area Under the Plasma Concentration-time Curve From Time 0 to Time Tau Over the Dosing Interval for TAK-906 and Its Metabolite M23 on Day 1 of Single Dose Period
Description: AUCtau is a measure of total plasma exposure to TAK-906 and its Metabolite M23 from Time 0 to Time tau over the dosing interval.
Time Frame: Day 1 pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours post-dose
Population: as for outcome 6
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Cohort 1: TAK-906 50 mg | Cohort 2: TAK-906 100 mg | Cohort 3: TAK-906 10 mg
Number analyzed (Participants) | 6 | 6 | 6
h*ng/mL
  TAK-906 | 70.96 (16.586) | 149.1 (39.145) | 13.47 (2.0130)
  Metabolite M23 | 7.608 (1.8894) | 14.69 (6.8520) | 1.327 (0.60977)

9. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-906 and Its Metabolite M23 on Day 1 of Single Dose Period
Description: Tmax is time to reach the peak plasma concentration of TAK-906 and its metabolite M23.
Time Frame: Day 1 pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours post-dose
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1: TAK-906 50 mg | Cohort 2: TAK-906 100 mg | Cohort 3: TAK-906 10 mg
Number analyzed (Participants) | 6 | 6 | 6
hours
  TAK-906 | 1.000 [1.00 to 2.00] | 1.000 [0.500 to 3.00] | 1.000 [1.00 to 1.50]
  Metabolite M23 | 1.000 [1.00 to 2.00] | 1.000 [1.00 to 4.00] | 1.000 [1.00 to 1.50]

10. Secondary Outcome: t1/2z: Terminal Disposition Phase Half-life for TAK-906 and Its Metabolite M23 on Day 1 of Single Dose Period
Description: t1/2z is time for the plasma concentration of TAK-906 and its metabolite M23 to decrease by half.
Time Frame: Day 1 pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1: TAK-906 50 mg | Cohort 2: TAK-906 100 mg | Cohort 3: TAK-906 10 mg
Number analyzed (Participants) | 6 | 6 | 6
hours
  TAK-906 | 4.692 (3.8389) | 5.152 (2.1478) | 1.894 (0.85198)
  Metabolite M23 | 2.483 (1.2160) | 4.423 (3.0935) | 3.170 (2.2826)

11. Secondary Outcome: Ae(0-24): Amount of Drug Excreted in Urine From Time 0 to 24 Hours Postdose for TAK-906 and Its Metabolite M23 on Day 1 of Single Dose Period
Description: Ae(0-24) is the amount of TAK-906 and its metabolite M23 excreted in urine from Time 0 to 24 Hours postdose.
Time Frame: Day 1 pre-dose and 0-6, 6-12, and 12-24 hours post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: microgram (mcg)
Arm/Group | Cohort 1: TAK-906 50 mg | Cohort 2: TAK-906 100 mg | Cohort 3: TAK-906 10 mg
Number analyzed (Participants) | 6 | 6 | 6
microgram (mcg)
  TAK-906 | 741.2 (114.12) | 1571 (621.57) | 160.0 (29.766)
  Metabolite M23 | 64.57 (23.741) | 135.2 (80.915) | 13.27 (6.5007)

12. Secondary Outcome: Fe24: Fraction of Administered Dose of Drug Excreted in Urine From Time 0 to 24 Hours for TAK-906 and Its Metabolite M23 on Day 1 of Single Dose
Description: Fe24 was calculated as percentage of administered dose of drug excreted in urine from Time 0 to 24 Hours for TAK-906 and its metabolite M23.
Time Frame: Time Frame Day 1 pre-dose and 0-6, 6-12, and 12-24 hours post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percentage of drug
Arm/Group | Cohort 1: TAK-906 50 mg | Cohort 2: TAK-906 100 mg | Cohort 3: TAK-906 10 mg
Number analyzed (Participants) | 6 | 6 | 6
percentage of drug
  TAK-906 | 1.815 (0.27941) | 1.923 (0.76094) | 1.959 (0.36440)
  Metabolite M23 | 0.1575 (0.057901) | 0.1648 (0.098672) | 0.1618 (0.079274)

13. Secondary Outcome: CLR: Renal Clearance for TAK-906 and Its Metabolite M23 on Day 1 of Single Dose Period
Description: Renal clearance is a measure of apparent clearance of TAK-906 and its metabolite M23 from the urine.
Time Frame: Day 1 pre-dose and 0-6, 6-12, and 12-24 hours post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: liter per hour (L/h)
Arm/Group | Cohort 1: TAK-906 50 mg | Cohort 2: TAK-906 100 mg | Cohort 3: TAK-906 10 mg
Number analyzed (Participants) | 6 | 6 | 6
liter per hour (L/h)
  TAK-906 | 10.31 (1.9096) | 9.741 (2.5812) | 11.76 (2.4737)
  Metabolite M23 | 8.021 (1.6016) | 7.782 (2.0366) | 9.204 (2.8328)

14. Secondary Outcome: AUC(τ,ss): Area Under the Plasma Concentration-time Curve From Time 0 During Dosing Interval at Steady State for TAK-906 and Its Metabolite M23 on Day 7 of Multiple Dose Period
Description: AUC(τ,ss) is a measure of total plasma exposure to TAK-906 and its metabolite M23 from Time 0 during dosing interval at steady state.
Time Frame: Day 7 pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours post-dose
Population: as for outcome 6
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Cohort 1: TAK-906 50 mg | Cohort 2: TAK-906 100 mg | Cohort 3: TAK-906 10 mg
Number analyzed (Participants) | 6 | 6 | 6
h*ng/mL
  TAK-906 | 89.01 (9.0816) | 186.6 (9.5795) | 16.28 (1.6646)
  Metabolite M23 | 9.881 (2.7666) | 25.35 (9.4350) | 1.672 (0.48714)

15. Secondary Outcome: Cmax,ss: Maximum Observed Plasma Concentration During Dosing Interval at Steady State for TAK-906 and Its Metabolite M23 on Day 7 of Multiple Dose Period
Description: Cmax, ss is the peak plasma concentration of TAK-906 and its metabolite M23 during dosing interval at steady state.
Time Frame: Day 7 pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours post-dose
Population: as for outcome 6
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: TAK-906 50 mg | Cohort 2: TAK-906 100 mg | Cohort 3: TAK-906 10 mg
Number analyzed (Participants) | 6 | 6 | 6
ng/mL
  TAK-906 | 46.47 (12.173) | 79.36 (19.958) | 7.642 (2.8630)
  Metabolite M23 | 3.858 (2.2739) | 8.119 (4.0837) | 0.5309 (0.24586)

16. Secondary Outcome: Tmax,ss: Time to Reach the Maximum Plasma Concentration (Cmax) at Steady State for TAK-906 and Its Metabolite M23 on Day 7 of Multiple Dose Period
Description: Tmax,ss is defined as time to reach the peak plasma concentration at steady state for TAK-906 and its metabolite M23.
Time Frame: Day 7 pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours post-dose
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1: TAK-906 50 mg | Cohort 2: TAK-906 100 mg | Cohort 3: TAK-906 10 mg
Number analyzed (Participants) | 6 | 6 | 6
hours
  TAK-906 | 1.000 [0.500 to 1.50] | 1.250 [1.00 to 2.00] | 1.000 [0.500 to 1.00]
  Metabolite M23 | 1.000 [0.500 to 1.50] | 1.500 [1.00 to 2.00] | 1.000 [1.00 to 1.50]

17. Secondary Outcome: t1/2z: Terminal Disposition Phase Half-life for TAK-906 and Its Metabolite M23 on Day 7 of Multiple Dose Period
Description: t1/2z is time for the plasma concentration of TAK-906 and its metabolite M23 to decrease by half.
Time Frame: Day 7 pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Cohort 1: TAK-906 50 mg | Cohort 2: TAK-906 100 mg | Cohort 3: TAK-906 10 mg
Number analyzed (Participants) | 6 | 6 | 6
hour
  TAK-906 | 6.447 (2.4506) | 4.407 (1.1057) | 3.727 (2.9253)
  Metabolite M23 | 5.573 (2.7810) | 4.598 (0.85968) | 3.037 (2.8804)

18. Secondary Outcome: Aetau: Amount of Drug Excreted in Urine During a Dosing Interval for TAK-906 and Its Metabolite M23 on Day 7 of Multiple Dose Period
Description: Aetau is the amount of TAK-906 and its metabolite M23 excreted in urine during a dosing Interval.
Time Frame: Day 7 pre-dose and 0-6 and 6-12 hours post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | Cohort 1: TAK-906 50 mg | Cohort 2: TAK-906 100 mg | Cohort 3: TAK-906 10 mg
Number analyzed (Participants) | 6 | 6 | 6
mcg
  TAK-906 | 895.8 (179.72) | 2155 (358.71) | 198.7 (28.140)
  Metabolite M23 | 78.75 (29.365) | 237.7 (109.04) | 16.11 (7.2989)

19. Secondary Outcome: Fetau: Fraction of Administered Dose of Drug Excreted in Urine From Time 0 to Time Tau Over the Dosing Interval for TAK-906 and Its Metabolite M23 on Day 7 of Multiple Dose Period
Description: Fetau was calculated as percentage of administered dose of drug excreted in urine from Time 0 to Time tau over the dosing interval for TAK-906 and its metabolite M23.
Time Frame: Day 7 pre-dose and 0-6 and 6-12 hours post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percentage of drug
Arm/Group | Cohort 1: TAK-906 50 mg | Cohort 2: TAK-906 100 mg | Cohort 3: TAK-906 10 mg
Number analyzed (Participants) | 6 | 6 | 6
percentage of drug
  TAK-906 | 2.193 (0.44004) | 2.638 (0.43913) | 2.432 (0.34450)
  Metabolite M23 | 0.1921 (0.071618) | 0.2898 (0.13297) | 0.1965 (0.089007)

20. Secondary Outcome: CLR: Renal Clearance for TAK-906 and Its Metabolite M23 on Day 7 of Multiple Dose Period
Description: Renal clearance is a measure of apparent clearance of TAK-906 and its metabolite M23 from the urine.
Time Frame: Day 7 pre-dose and 0-6 and 6-12 hours post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Cohort 1: TAK-906 50 mg | Cohort 2: TAK-906 100 mg | Cohort 3: TAK-906 10 mg
Number analyzed (Participants) | 6 | 6 | 6
L/h
  TAK-906 | 10.04 (1.8881) | 11.50 (1.5423) | 12.21 (1.7620)
  Metabolite M23 | 7.744 (1.6110) | 8.669 (0.99318) | 9.113 (2.2294)

21. Secondary Outcome: AUCtau: Area Under the Serum Concentration-time Curve During a Dosing Interval for Serum Prolactin on Day 1 of Single Dose Period
Description: AUCtau defined as area under the serum concentration-time curve during a dosing interval for serum prolactin was calculated.
Time Frame: Day 1 pre-dose and 1, 2, 4, 6, and 24 hours post-dose
Population: The pharmacodynamics (PD) analysis set consisted of participants who received at least 1 dose of study drug, completed the minimum protocol-specified procedures with no significant protocol deviations, and who were evaluable for the PD.
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Cohorts 1-3: Placebo | Cohort 1: TAK-906 50 mg | Cohort 2: TAK-906 100 mg | Cohort 3: TAK-906 10 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
h*ng/mL | 79.66 (12.529) | 362.9 (101.53) | 398.7 (151.86) | 317.4 (136.71)

22. Secondary Outcome: Cmax: Maximum Observed Serum Concentration for Serum Prolactin on Day 1 of Single Dose Period
Description: Cmax is the peak serum concentration of serum prolactin.
Time Frame: Day 1 pre-dose and 1, 2, 4, 6, and 24 hours post-dose
Population: The PD analysis set consisted of participants who received at least 1 dose of study drug, completed the minimum protocol-specified procedures with no significant protocol deviations, and who were evaluable for the PD.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohorts 1-3: Placebo | Cohort 1: TAK-906 50 mg | Cohort 2: TAK-906 100 mg | Cohort 3: TAK-906 10 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng/mL | 10.68 (1.9500) | 73.12 (37.398) | 81.09 (55.593) | 82.33 (45.405)

23. Secondary Outcome: AUClast: Area Under the Serum Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Serum Prolactin on Day 1 of Single Dose Period
Description: AUClast defined as area under the serum concentration-time curve from Time 0 to the Time of the last quantifiable concentration for serum prolactin was calculated.
Time Frame: Day 1 pre-dose and 1, 2, 4, 6, and 24 hours post-dose
Population: as for outcome 22
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Cohorts 1-3: Placebo | Cohort 1: TAK-906 50 mg | Cohort 2: TAK-906 100 mg | Cohort 3: TAK-906 10 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
h*ng/mL | 174.5 (26.584) | 544.9 (120.83) | 638.8 (171.24) | 449.9 (167.52)

24. Secondary Outcome: AUC(t,ss): Area Under the Serum Concentration-time Curve From Time 0 During Dosing Interval at Steady State for Serum Prolactin on Day 7 of Multiple Dose Period
Description: AUC(t,ss) defined as area under the serum concentration-time curve from Time 0 during dosing interval at steady state for serum prolactin was calculated.
Time Frame: Day 7 pre-dose and 1, 2, 4, 6, and 24 hours post-dose
Population: as for outcome 22
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Cohorts 1-3: Placebo | Cohort 1: TAK-906 50 mg | Cohort 2: TAK-906 100 mg | Cohort 3: TAK-906 10 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
h*ng/mL | 75.40 (9.8027) | 354.8 (142.68) | 476.2 (122.05) | 317.0 (147.70)

25. Secondary Outcome: Cmax,ss: Maximum Observed Serum Concentration During Dosing Interval at Steady State for Serum Prolactin on Day 7 of Multiple Dose Period
Description: Cmax,ss is the peak serum concentration of serum prolactin during dosing interval at steady state.
Time Frame: Day 7 pre-dose and 1, 2, 4, 6, and 24 hours post-dose
Population: as for outcome 22
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohorts 1-3: Placebo | Cohort 1: TAK-906 50 mg | Cohort 2: TAK-906 100 mg | Cohort 3: TAK-906 10 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng/mL | 11.48 (3.4891) | 39.65 (16.014) | 55.89 (20.890) | 71.02 (38.025)

ADVERSE EVENTS:
Time Frame: TEAEs are adverse events that started after the first dose of double-blind study drug up to Day 14
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Cohorts 1-3: Placebo | Cohort 1: TAK-906 50 mg | Cohort 2: TAK-906 100 mg | Cohort 3: TAK-906 10 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/6 | 0/6 | 2/6 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohorts 1-3: Placebo (N=6) | Cohort 1: TAK-906 50 mg (N=6) | Cohort 2: TAK-906 100 mg (N=6) | Cohort 3: TAK-906 10 mg (N=6)
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2017-06-06): https://cdn.clinicaltrials.gov/large-docs/56/NCT03237156/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-10): https://cdn.clinicaltrials.gov/large-docs/56/NCT03237156/SAP_001.pdf